CLINICAL TRIAL: NCT03795012
Title: A Multicenter, Randomized, Phase II Trial Evaluating the Efficacy of Eribulin Monotherapy and Eribulin Plus Endocrine Therapy in Locally-recurrent or Metastatic Breast Cancer Patients After Progression on Endocrine Therapy (REVERT)
Brief Title: Trial With Eribulin or Eribulin+ Endocrine Therapy in Locally-recurrent or Metastatic Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP167; 2017-004324-30 (EudraCT Number)
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; Unresectable; ER; PR; Her2; recurrent; metastatic
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasm Metastasis | interventions — eribulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eribulin monotherapy (Active Comparator): Patients will receive eribulin injections intravenously on days 1 and 8 of every 21- day cycle
  Interventions: Drug: Eribulin
- eribulin plus endocrine therapy (Active Comparator): Patients will receive eribulin injections intravenously on days 1 and 8 of every 21- day cycle, in combination with endocrine therapy (aromatase inhibitor). AI must be identical to the last AI administered to the patient, whether in the adjuvant or metastatic setting.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — Patients will receive eribulin injections intravenously on days 1 and 8 of every 21-day cycle alone.
  Other Names: Halaven

SUMMARY:
Unresectable, ER-positive and/or PR-positive and HER2-negative locally-recurrent or metastatic breast cancer (mBC).

DETAILED DESCRIPTION:
Pre- and post-menopausal women age ≥ 18 years with unresectable, ER-positive and/or PR-positive and HER2-negative locally-recurrent or metastatic breast cancer (mBC) with no prior line of chemotherapy in the metastatic setting, and that have shown progression while on an aromatase inhibitor-containing regimen in the metastatic setting or within six months from last aromatase inhibitor dose in the adjuvant setting. Patients must have received at least one taxane or anthracycline regimen in either the adjuvant or the neoadjuvant setting. Subjects must have adequate bone marrow and creatinine clearance functions.

ELIGIBILITY:
Inclusion Criteria:

* ER-positive and/or PR-positive breast cancer.
* HER2-negative breast cancer.
* Unresectable locally advanced or metastatic breast cancer.
* Confirmed disease progression while in the last aromatase inhibition-containing regimen in the metastatic setting.
* At least one taxane or anthracycline regimen in either the adjuvant or the neoadjuvant setting.
* Patients with no prior line of chemotherapy in the metastatic setting.
* At least 1 and up to 3 prior lines of endocrine therapy in the metastatic setting.
* ECOG score 0 or 1.
* Patients have adequate bone marrow and organ function.
* Patients must have measurable disease (RECIST v.1.1).
* Premenopausal with LHRH analogues for at least 28 days) and postmenopausal women.
* Patients must agree to not breastfeed during the study and for 3 months after the last dose of study treatment.
* Life expectancy greater or equal to 12 weeks.
* Patients agree to collection of blood samples (liquid biopsy) and optional collection of metastatic tumour sample (biopsy) at the time of inclusion and progression (if appropriate).

Exclusion Criteria:

* Have received radiation therapy or limited-field palliative radiotherapy within two weeks prior to Cycle 1, Day 1, or patients who have not recovered from radiotherapy-related toxicities.
* Have received prior chemotherapy for locally advanced or metastatic disease.
* Have peripheral neuropathy grade 2 or greater.
* QTc > 480 msec on basal assessments, history of congenital or personal history of long QT syndrome, Brugada syndrome, or Torsade de Pointes (TdP), or uncontrolled electrolyte disorders
* Child-bearing potential women not using highly effective methods of contraception.
* Known hypersensitivity to eribulin, endocrine therapy or its excipients.
* Other malignancies within the previous two years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of cervix or breast.
* Known uncontrolled metastases to the central nervous system (CNS) or any progressing CNS disease.
* Have a serious concomitant systemic disorder incompatible with the study.
* Major surgical procedure or significant traumatic injury within 28 days prior to randomization.
* Have received any anti-cancer biology or investigational treatment within 30 days prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The overall response rate (ORR) | Baseline up to 27 months
  The overall response rate (ORR) in the eribulin + ET arms, defined as the proportion of patients with best overall response of confirmed complete response or partial response based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria v. 1.11.

SECONDARY OUTCOMES:
The progression-free survival (PFS) | Baseline up to 27 months
  The progression-free survival (PFS) for patients treated with endocrine therapy alone or in combination with eribulin is defined as the time from randomization until death by any cause or objective tumor progression based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria v. 1.11.
PFS-2, in the eribulin and the eribulin + ET arms | Baseline up to 27 months
  The PFS-2, in the eribulin and the eribulin + ET arms, defined as the time from the randomization to the second disease progression or death, i.e., PFS after the next line of treatment, based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria v. 1.11.
Overall response rate (ORR) in the eribulin arm | Baseline up to 27 months
  The overall response rate (ORR) in the eribulin arm, defined as the proportion of patients with best overall response of confirmed complete response or partial response based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria v. 1.11.
The duration of response (DOR) in the eribulin and the eribulin + ET arms | Baseline up to 27 months
  The duration of response (DOR) in the eribulin and the eribulin + ET arms, defined as the time from the start of the treatment to disease progression based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria v. 1.11.
The clinical benefit rate (CBR) in the eribulin and the eribulin + ET arms | Baseline up to 27 months
  The clinical benefit rate (CBR) in the eribulin and the eribulin + ET arms, defined as the proportion of patients with no disease progression after 6 months of therapy, based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria v. 1.11.
The overall survival (OS) in the eribulin and the eribulin + ET arms | Baseline up to 27 months
  The overall survival (OS) in the eribulin and the eribulin + ET arms, defined as the length of time that patients remain alive from the start of treatment (OS will be collected at the end of the study).
Maximum Tumor shrinkage | Baseline up to 27 months
  Maximum Tumor shrinkage, defined as the percentage of tumor shrinkage from baseline (obtained from the sum of the largest diameters of the target lesions), based on local investigator's assessment according to RECIST criteria guidelines (version 1.1)1.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, PhD, Principal Investigator — MedSIR
Locations (9):
- Spain (9):
  - Hospital de Jaén, Jaén, Jaén
  - Hospital Quiron Dexeus, Barcelona, Please Select
  - Institut Català d'Oncologia, Girona
  - Complejo Asistencial Universitario de León, León
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz,, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario Dr Peset, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No